CLINICAL TRIAL: NCT04770142
Title: The Study for Evaluation of Safety and Efficacy of Transcatheter RF Ablation System (TIRA Catheter) to Treat Hypertrophic Obstructive Cardiomyopathy : Multi-center, Open Label, Single Arm, Investigator Initiated Exploratory Pilot Study
Brief Title: First-in-Man Early Feasibility Study for Transcatheter HOCM Septal Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: During the course of the clinical trial, sufficient subject enrollment was not achieved. As the recruitment of additional subjects was considered practically unfeasible, the clinical trial was terminated early.
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seung-Whan Lee,MD,PhD, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TIRA-FIM
Record Dates: First submitted 2021-02-17; First posted 2021-02-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Transcatheter RF ablation; Intraseptal ablation; HOCM; TauPnu
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: multi-center, open label, single arm, investigator initiated exploratory pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TIRA (Experimental): treated with transcatheter RF ablation system (TIRA catheter with its supplemental devices)
  Interventions: Device: TIRA catheter

INTERVENTIONS:
Device: TIRA catheter — treat hypertrophic obstructive cardiomyopathy
  Other Names: CA10 and ohter 3 models

SUMMARY:
Transcatheter Intra-septal RF ablation system (TIRA catheter with its supplemental devices) to treat hypertrophic obstructive cardiomyopathy.

DETAILED DESCRIPTION:
The objective of this multi-center, open label, single arm, investigator initiated exploratory pilot study is to evaluation of safety and efficacy of transcatheter Intra-septal RF ablation system (TIRA catheter with its supplemental devices), in treating hypertrophic obstructive cardiomyopathy(HOCM).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 20 years or older
* NYHA(New York Heart Association) Class Ⅱ to Ⅳ in spite of optimal medical treatment. (For optimal medical treatment, β-blocker or diuretic such as calcium antagonists should be given for at least 3 months.)
* Patients with left ventricular effusion gradient (LVOT) greater than (1) 30 mmHg at rest or (2) at least 50 mmHg at physiological exercise/dobutamine administration/balsalva manuver. (The pressure difference due to the left ventricle drain must be the proximal mitral valve-septal contact by the systolic motion of mitral valve (SAM).)
* Patients who voluntarily decide to participate in this clinical trial and provide written informed consent.
* Patients who are able to understand and follow instructions and participate for the entire duration of the clinical trial.

Exclusion Criteria:

* Target area wall thickness ≤15mm
* LV ejection fraction ≤40%
* Subjects who have unsuitable septal vein and coronary sinus anatomy by cardiac CT or venogram
* Conduction disturbance; LBBB or RBBB
* Advanced AV block without permanent pacemaker
* Subjects who have experience in performing vascular stent procedures (PCI) or CABG on coronary arteries close to the coronary sinus within 3 months.
* Severe pulmonary HTN ≥70mmHg
* Patients who have cardiogenic shock and those who have an expected life expectancy of 12 months or less.
* Patients with other valve diseases (companion disease) that require surgical treatment (in this case, Systolic motion of the mitral valve (SAM) caused by systolic myocardia is not considered a companion disease).
* Patients who are pregnant, or lactating, or plan pregnacy during the clinical trials
* Patients who are participated in other clinical trials within 1 month of enrollment
* Patients who are deemed not to be eligible in this study by physician's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change of LVOT obstruction | immediately after the procedure and 3 months
  LVOT gradient (mmHg) ; resting / valsalva maneuver with Echocardiogram
Change of LVOT and Septum(1) | immediately after the procedure and 3 months
  LVOT diameter (mm) with Echocardiogram
Change of LVOT and Septum(2) | immediately after the procedure and 3 months
  Intraventricular septum(IVS) thickness (mm) with Echocardiogram
Morphological Structural Changes in the Lesion Area | immediately after the procedure and 3 months
  Intraventricular septum(IVS) thickness (mm) with cardiac CT and MRI
Rate of adverse events as a measure of safety | immediately after the procedure and 3 months
  Adverse Events (AEs): Frequency (Number of Events)
  *with particular focus on serious adverse events (SAEs) and serious adverse device effects (SADEs).

SECONDARY OUTCOMES:
Change of LVOT obstruction | 6 and 12 months
  LVOT gradient (mmHg) ; resting / valsalva maneuver with Echocardiogram
Change of LVOT and Septum(1) | 6 and 12 months
  LVOT diameter (mm) with Echocardiogram
Change of LVOT and Septum(2) | 6 and 12 months
  Intraventricular septum(IVS) thickness (mm) with Echocardiogram
Change of LVOT and Septum(3) | 6 and 12 months
  Left atrial volume index (ml/m2) with Echocardiogram
Change of LVOT and Septum(4) | 6 and 12 months
  Mitral regurgitation volume (ml) with Echocardiogram
Change of LVOT and Septum(5) | 6 and 12 months
  Systolic anterior motion of the mitral valve (SAM) with Echocardiogram
Morphological Structural Changes in the Lesion Area | 6 and 12 months
  Intraventricular septum(IVS) thickness (mm) with cardiac CT and MRI
Rate of adverse events as a measure of safety | 6 and 12 months
  Adverse Events (AEs): Frequency (Number of Events)
  *with particular focus on serious adverse events (SAEs) and serious adverse device effects (SADEs).

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (9):
- South Korea (9):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Hallym University Medical Center, Anyang, Dongan-gu
  - Sejong HOSPITAL, Bucheon-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungnam National University Hospital (CNU Hospital), Daejeon, Jung-gu
  - Yeungnam University Hospital, Daegu, Nam-gu
  - Ulsan Hospital, Ulsan, Nam-gu
  - Chungnam National University Sejong Hospital, Sejong, Sejong-si
  - Asan Medical Center, Seoul, Songpa-gu

REFERENCES:
- [Background] Oh JS, Seo JY, Lee CM, Jung SJ, Kim JH, Chon MK. Trans-Coronary Sinus Intra-Septal Radiofrequency Ablation (TIRA) for Hypertrophic Obstructive Cardiomyopathy: First-in-Human Results. Biomedicines. 2024 Dec 4;12(12):2762. doi: 10.3390/biomedicines12122762. PMID 39767669